CLINICAL TRIAL: NCT04002531
Title: A One Visit Follow Up of Adults With Fabry Disease Who Started Long-term Enzyme Replacement Therapy As Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Baylor Research Institute (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 018-706
Record Dates: First submitted 2019-03-25; First posted 2019-06-28 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-03

CONDITIONS: Quality of Life; Renal Insufficiency; Cardiac Event
MeSH Terms: conditions — Renal Insufficiency; Cardiovascular Diseases | interventions — Blood Pressure; Heart Rate; Respiratory Rate; epicatechin gallate; Blood Specimen Collection; Phlebotomy; Urine Specimen Collection; bactericidal permeability increasing protein

STUDY DESIGN:
Intervention Model Description: Specific group of adults with Fabry disease who received Replagal infusions as children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Visit (Other): 1. General and neurological examination
  2. Vital signs including height, weight, blood pressure, pulse, temperature
  3. 12 lead ECG
  4. 2 hour Holter monitor for heart rate variability
  5. Echocardiogram
  6. Renal function will be assessed by the eGFR. The eGFR will be calculated from serum creatinine using CKD-EPI equation.
  7. CBC with differential
  8. Complete metabolic panel
  9. Urinalysis
  10. Urine Albumin/creatinine ratio.
  11. Urine and plasma samples for biomarkers (Gb3, lyso-Gb3) that will be stored in -80 freezer and assayed in our lab.
  12. Brief Pain Inventory questionnaire.
  13. Quality of Life Questionnaires (SF36)
  Interventions: Other: General and Neurological examination; Other: Vital signs; Procedure: 12 lead electrocardiogram; Procedure: Echocardiogram; Procedure: Blood draw; Procedure: Urine collection; Procedure: 2-hour Holter Monitor; Other: Brief Pain Inventory questionnaire; Other: Quality of Life questionnaire

INTERVENTIONS:
Other: General and Neurological examination — Information about your general health, neurological symptoms and current medications with be collected
  Other Names: MD assessment
Other: Vital signs — Height, weight, blood pressure, heart rate, and respiratory rate and temperature will be measured.
  Other Names: Blood pressure, heart rate, respiratory rate
Procedure: 12 lead electrocardiogram — A non-invasive test that measures the electrical activity of the heart
  Other Names: EKG, ECG
Procedure: Echocardiogram — A non-invasive sonogram of the heart
  Other Names: Cardiac echo
Procedure: Blood draw — Blood will be drawn to evaluate general health and renal function (kidney health)
  Other Names: Blood collection, phlebotomy, lab test
Procedure: Urine collection — Urine will be collection to evaluate renal function (kidney health)
Procedure: 2-hour Holter Monitor — A non-invasive test that measures the electrical activity of the heart continuously over 2 hours
  Other Names: Holter
Other: Brief Pain Inventory questionnaire — A questionnaire about daily pain
  Other Names: BPI, Pain questionnaire
Other: Quality of Life questionnaire — A questionnaire about the impact of disease on their activities of daily living and quality of life
  Other Names: SF 36

SUMMARY:
The objective of this study is to obtain follow up data on a cohort of well-studied patients with Fabry disease who have been on ERT since childhood for a total of about 15 years.

DETAILED DESCRIPTION:
The long-term effect of initiating ERT in childhood is unknown. Prospective studies of Children with Fabry disease on 0.2 mg/kg agalsidase alfa every other week were performed. The patients were 7-17 years of age at initial study enrollment. The first open-label protocol was TKT023, a 6 months study (August 12, 2002-October 20, 2004) that was followed by an extension study TKT029 (June 10, 2004-June 15, 2011; ClinicalTrials.gov identifier NCT00084084). Since completing TKT029, all US patients were switched to commercial agalsidase beta. Therefore, these patients have now been treated for about 15 years.This study involves a one-visit follow up on these patients using the same protocol-driven studies as were used in TKT029. The long-term follow up data gathered will consist of a rare description of the disease profile in patients who were treated with ERT since childhood.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who participated in TKT029 and who are willing and able to come to Dallas for 1 visit for standard of care testing.
2. Sign the protocol informed consent form
3. Have been on continuous commercial ERT since TKT029 has ended

Exclusion Criteria:

1. Patients who are unable to understand the nature, scope, and possible consequences of the study.
2. Patient does not give his written informed consent to participate in this study
3. Patient is unable to comply with the protocol, e.g., uncooperative with protocol schedule, refusal to agree to all of the study procedures.
4. Patient has been off ERT for an extended period of time as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
estimated Glomerular Filtration Rate (eGFR) | Study involves one visit only - assessed Baseline Visit
  Change in eGFR since previous participation in study "Replagal Enzyme Replacement Therapy for Children With Fabry Disease" - NCT00084084

SECONDARY OUTCOMES:
Left Ventricular Mass Index | Study involves one visit only - assessed Baseline Visit
  LVMI measured in g/m2 by echocardiogram and compared to LVMI results obtained during participation in study "Replagal Enzyme Replacement Therapy for Children With Fabry Disease" NCT00084084
Heart rate variability assessment | Study involves one visit only - assessed Baseline Visit
  2 hour holter monitor and compared to holter monitor results obtained during participation in study "Replagal Enzyme Replacement Therapy for Children With Fabry Disease" NCT00084084
Urine albumin/creatinine ratio | Study involves one visit only - assessed Baseline Visit
  Biomarker of renal function and compared to urine albumin/creatinine ratios obtained during participation in study "Replagal Enzyme Replacement Therapy for Children With Fabry Disease" NCT00084084
Plasma Lyso-Gb3 | Study involves one visit only - assessed Baseline Visit
  Biomarker of disease and compared to plasma Lyso-Gb3 results obtained during participation in study "Replagal Enzyme Replacement Therapy for Children With Fabry Disease" NCT00084084
Plasma Gb3 and compared to plasma Gb3 results obtained during participation in study "Replagal Enzyme Replacement Therapy for Children With Fabry Disease" NCT00084084 | Study involves one visit only - assessed Baseline Visit
  Biomarker of disease
Urine Lyso-Gb3 | Study involves one visit only - assessed Baseline Visit
  Biomarker of disease and compared to urine Lyso-Gb3 results obtained during participation in study "Replagal Enzyme Replacement Therapy for Children With Fabry Disease" NCT00084084
Short-form Brief Pain Inventory (BPI) | Study involves one visit only - assessed Baseline Visit
  Questionnaire designed to assess current level of pain from 0-10. 0 reflects no pain and 10 being the worst possible pain. Results will be compared to pediatric pain assessments obtained during participation in study "Replagal Enzyme Replacement Therapy for Children With Fabry Disease" NCT00084084
Qualify of Life - Your Health and Well-being | Study involves one visit only - assessed Baseline Visit
  Self-evaluation that describes current physical and emotional health. Questionnaire asks User to rate how Fabry disease impacts User's overall physical and emotional well-being. Questionnaire uses multiple scales to rate User's ability to perform activities of daily life, identify changes in overall health, and identify how changes in physical health and disease has impacted User's emotional well-being. User will be asked to answer multiple questions using the following scales: Poor/Fair/Good/Very good/excellent, Much better than 1 week ago/Somewhat better than 1 week ago/The same as 1 week ago/Somewhat worse than 1 week ago/Much worse than 1 week ago, Limited a lot/Limited a little/Not limited at all, All of the time/Most of the time/Some of the time/A little of the time/None of the time, Not at all/Slightly/Moderately/Quite a bit/Extremely, None/Very mild/Mild/Moderate/Severe/Very severe, Definitely true/Mostly true/Don't know/Mostly false/Definitely false.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schiffmann R. Fabry disease. Pharmacol Ther. 2009 Apr;122(1):65-77. doi: 10.1016/j.pharmthera.2009.01.003. Epub 2009 Feb 8. PMID 19318041
- [Background] Schiffmann R, Ries M. Fabry Disease: A Disorder of Childhood Onset. Pediatr Neurol. 2016 Nov;64:10-20. doi: 10.1016/j.pediatrneurol.2016.07.001. Epub 2016 Jul 29. PMID 27555236
- [Background] Echevarria L, Benistan K, Toussaint A, Dubourg O, Hagege AA, Eladari D, Jabbour F, Beldjord C, De Mazancourt P, Germain DP. X-chromosome inactivation in female patients with Fabry disease. Clin Genet. 2016 Jan;89(1):44-54. doi: 10.1111/cge.12613. Epub 2015 Jun 22. PMID 25974833
- [Background] Dobyns WB. The pattern of inheritance of X-linked traits is not dominant or recessive, just X-linked. Acta Paediatr Suppl. 2006 Apr;95(451):11-5. doi: 10.1111/j.1651-2227.2006.tb02383.x. PMID 16720459
- [Background] MacDermot KD, Holmes A, Miners AH. Natural history of Fabry disease in affected males and obligate carrier females. J Inherit Metab Dis. 2001;24 Suppl 2:13-4; discussion 11-2. doi: 10.1023/a:1012447102358. No abstract available. PMID 11758673
- [Background] Schiffmann R, Warnock DG, Banikazemi M, Bultas J, Linthorst GE, Packman S, Sorensen SA, Wilcox WR, Desnick RJ. Fabry disease: progression of nephropathy, and prevalence of cardiac and cerebrovascular events before enzyme replacement therapy. Nephrol Dial Transplant. 2009 Jul;24(7):2102-11. doi: 10.1093/ndt/gfp031. Epub 2009 Feb 13. PMID 19218538
- [Background] Kwon JM, Matern D, Kurtzberg J, Wrabetz L, Gelb MH, Wenger DA, Ficicioglu C, Waldman AT, Burton BK, Hopkins PV, Orsini JJ. Consensus guidelines for newborn screening, diagnosis and treatment of infantile Krabbe disease. Orphanet J Rare Dis. 2018 Feb 1;13(1):30. doi: 10.1186/s13023-018-0766-x. PMID 29391017
- [Background] Meikle PJ, Hopwood JJ, Clague AE, Carey WF. Prevalence of lysosomal storage disorders. JAMA. 1999 Jan 20;281(3):249-54. doi: 10.1001/jama.281.3.249. PMID 9918480
- [Background] Schiffmann R, Hughes DA, Linthorst GE, Ortiz A, Svarstad E, Warnock DG, West ML, Wanner C; Conference Participants. Screening, diagnosis, and management of patients with Fabry disease: conclusions from a "Kidney Disease: Improving Global Outcomes" (KDIGO) Controversies Conference. Kidney Int. 2017 Feb;91(2):284-293. doi: 10.1016/j.kint.2016.10.004. Epub 2016 Dec 18. PMID 27998644
- [Background] Schiffmann R, Pastores GM, Lien YH, Castaneda V, Chang P, Martin R, Wijatyk A. Agalsidase alfa in pediatric patients with Fabry disease: a 6.5-year open-label follow-up study. Orphanet J Rare Dis. 2014 Nov 26;9:169. doi: 10.1186/s13023-014-0169-6. PMID 25425121
- See also: Is it Fabry Disease? — https://www.nature.com/articles/gim201655